CLINICAL TRIAL: NCT05114434
Title: EFfect of FIxed Triple Beclometasone/Formoterol/Glycopyrronium Therapy on Cough effiCAcy in Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD) patiEnts: EFFICACE
Brief Title: Effect of BDP/Formoterol/G on Cough Efficacy in Moderate to Severe COPD Patients (EFFICACE)
Acronym: EFFICACE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Parma (Other)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: 38097
Record Dates: First submitted 2021-10-05; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: COPD, Chronic Obstructive Pulmonary Disease
Keywords: COPD; Beclometasone/Formoterol/Glycopyrronium (BDP/F/G); Cough Peak Flow (CPF)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective, single centre, 8 weeks, open-label study is designed to evaluate in real-life the effect of triple Beclometasone/Formoterol/Glycopyrronium (BDP/F/G) therapy on cough efficacy, assessed by cough peak flow (CPF), after 8 weeks' treatment in patients with moderate to severe COPD.

The study's hypothesis is that in symptomatic moderate to severe COPD patients the administration of fixed dose combination BDP/F/G, by reducing lung hyperinflation (LH) and targeting small airways, may accordingly improve the cough efficacy. The increase in cough efficacy might in turn positively influence the quality of life of patients and underlie the prevention of acute exacerbations of COPD.

DETAILED DESCRIPTION:
The cough is a vital defensive mechanism of respiratory system. Chronic obstructive pulmonary disease (COPD) is characterised by persistent inflammation in the small airways inducing pathological changes that reduce airflow and increase gas trapping and lung hyperinflation (LH). LH in turn leads to the changes in diaphragmatic excursions: this might decrease the efficacy of cough. In moderate to severe COPD patients, the cough efficacy, expressed as cough peak flow (CPF) and cough expired volume (CEV), is significantly reduced when compared to those of controls.

A triple combination inhaler containing beclometasone dipropionate/formoterol/glycopyrronium (BDP/F/G) was developed as an extrafine formulation to enable efficient delivery of an inhaled corticosteroid (ICS) combined with a long-acting beta2 agonist (LABA) and a long-acting muscarinic antagonist (LAMA) to the small airways, improving LH and associated symptoms.

The study's hypothesis is that the administration of fixed extrafine BDP/F/G 87/5/9 µg q.d. for 8 weeks will determine an increase of CPF, CEV, lung function and quality of life in COPD patients non adequately controlled by double combination of inhaled treatment with ICS plus LABA or ICS plus LAMA or LABA plus LAMA.

CPF, CEV, residual volume (RV), inspiratory capacity (IC), total lung capacity (TLC), RV/TLC ratio, forced expiratory volume at 1st second (FEV1), forced vital capacity (FVC) and FEV1/FVC ratio will be assessed at baseline (Visit 1, V1) and after 4 weeks' treatment with BDP/F/G (Visit 2, V2). The same assessments will be performed after 4 weeks' treatment (Visit 3, V3).

The switch from the double to triple therapy will be carried out according to clinical practice and to the summary of product characteristics.

At V1, V2, and V3 dyspnoea perception, assessed by the modified Medical Research Council (mMRC) scale score and the quality of life, assessed by the COPD Assessment Test (CAT), will be recorded.

V1, V2, V3 will be performed in the morning between 8:00 and 10:00 ante meridien.

Each patient will sign an informed consent prior to initiation of any study-related procedure. The study protocol was approved by the local Hospital's Ethical Committee (approval number n. 38097; September 22, 2021) and it will be conducted according to the Good Clinical Practices and the Declaration of Helsinki.

The population will consist of 40 adult patients. Assuming a p values < 0.05, a sample size of 40 patients (34 + 15% drop outs) is required to detect difference of 0.4 L/s (liters/second) with a standard deviation (SD) of 0.69 in CPF following a 8 weeks BDP/F/G treatment, with a power of 90%. Efficacy endpoints will be analysed using the intention to treat analysis (ITT) which will comprise all patients treated for 8 weeks with BDP/F/G 87/5/9 µg q.d. at visit 3.

Data will be collected in a dedicated electronic Clinical Records Form (CRF). The database will be saved on a password-protected company Personal Computer (PC) which will be updated at each visit and used exclusively for scientific research purposes. At the time of enrollment, each patient will receive an alphanumeric code so that any information collected during the study, and in particular sensitive data, is treated in an anonymous manner. Data reporting patients' identifications will only be used to file patients and collect informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged ≥40 years;
* Signed informed consent;
* Current or ex-smokers with a smoking history of at least 10 pack years. An ex smoker will be defined as a subject who has not smoked for ≥ 6months at screening;
* Diagnosis of COPD according to the International Statement;
* COPD patients with a forced expiratory volume in the 1st second (FEV1) between 30% and 80% of predicted post-bronchodilator (salbutamol 400 µg) at baseline visit;
* COPD patients with lung hyperinflation with residual volume (RV) ≥ 120% predicted;
* COPD patients treated with ICS/LABA or LABA/LAMA or ICS/LAMA therapy from at least one month before baseline visit;
* COPD patients with elevated impact of disease and/or symptoms defined by a CAT≥ 10 score and/or a mMRC ≥ 2 score and an history of exacerbation (≥ 1 exacerbation in the previous year).

Exclusion Criteria:

* Patients with COPD exacerbation that required treatment with antibiotics, systemic steroids (oral or intravenous) or hospitalization in the 4 weeks prior to enrolment;
* Patients with concomitant other lung disease (e.g. asthma, lung fibrosis, primary bronchiectasis, sarcoidosis, interstitial lung disorder, pulmonary hypertension);
* Patients requiring long-term oxygen therapy (LTOT) ≥12 h a day on a daily basis for chronic hypoxemia;
* Patients with severe comorbidities associated to COPD, such as unstable cardiovascular diseases or cancer;
* Patients with narrow-angle glaucoma, symptomatic benign prostatic hyperplasia (BPH), bladder-neck obstruction, moderate to severe renal impairment or urinary retention. BPH patients who are stable on treatment will be considered for enrolment;
* Patients with clinically significant renal, cardiovascular (such as but not limited to unstable ischemic heart disease, New York Heart Association (NYHA) Class III/IV left ventricular failure, myocardial infarction), neurological, endocrine, immunological, psychiatric, gastrointestinal, hepatic, or haematological abnormalities which could interfere with the assessment of the efficacy and safety of the study treatment;
* COPD patients treated with triple LABA/LAMA/ICS therapy;
* Pregnant women;
* Subjects unable to meet the criteria of acceptability and repeatability of pulmonary function tests, according to the American Thoracic Society/European Respiratory Society (ATS/ERS) document.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will consist of 40 adult patients, referred at outpatient clinic of the Respiratory Disease Unit of the University Hospital of Parma (Italy)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of fixed triple therapy BDP/F/G 87/5/9 μg q.d on cough efficacy after 8 weeks' treatment in moderate to severe COPD patients. | 8 weeks (4 weeks from V1 to V2; 4 weeks from V2 to V3)
  Increase of Cough Peak Flow (CPF, L/s) between V2 and V1 (Δ1) and from V3 and V2 (Δ2) will be compared as primary endpoint; superiority will be investigated comparing CPF values Δ2 versus Δ1.

SECONDARY OUTCOMES:
To evaluate the effect of the increase of CPF after 8 weeks' treatment with BDP/F/G on the cough expired volume. | 8 weeks (4 weeks from V1 to V2; 4 weeks from V2 to V3)
  Evaluation of changes between V2 and V1 (Δ1) and from V3 to V2 (Δ2) in Cough Expired Volume (CEV) (Liters, L).
To evaluate the effect of the increase of CPF after 8 weeks' treatment with BDP/F/G on dynamic lung volumes. | 8 weeks (4 weeks from V1 to V2; 4 weeks from V2 to V3)
  Improvement Δ1 and Δ2 in lung function assessed by means of spirometry parameters: Forced Expired Volume at 1 second (FEV1) (liters, L) and Forced Vital Capacity (FVC) (liters, L).
To evaluate the effect of the increase of CPF after 8 weeks' treatment with BDP/F/G on the airflow obstruction. | 8 weeks (4 weeks from V1 to V2; 4 weeks from V2 to V3)
  Improvement Δ1 and Δ2 in the index of airflow obstruction: Forced Expired Volume at 1 second (FEV1)/Forced Vital Capacity (FEV1/FVC) (%), assessed by means of spirometry.
To evaluate the effect of the increase of CPF after 8 weeks' treatment with BDP/F/G on static lung volumes, pulmonary capacity and lung hyperinflation. | 8 weeks (4 weeks from V1 to V2; 4 weeks from V2 to V3)
  Improvement Δ1 and Δ2 in plethysmograph parameters: Residual Volume (RV) (liters, L); Inspiratory Capacity (IC) (liters, L); Total Lung Capacity (TLC) (liters, L).
To evaluate the effect of the increase of CPF after 8 weeks' treatment with BDP/F/G on small airways dysfunction. | 8 weeks (4 weeks from V1 to V2; 4 weeks from V2 to V3)
  Improvement Δ1 and Δ2 in Impulse Oscillometry System (IOS) parameters: R5, Total resistance at 5 Hertz (Hz), KiloPascal/(L/s); R20, Central airway resistance at 20 Hz, KiloPascal/(L/s); R5-R20, fall in resistance from 5 Hz to 20 Hz, KiloPascal/(L/s) as index of peripheral (small) airways resistance; X5, reactance at 5 Hz, KiloPascal/(L/s).
To evaluate the effect of the increase of CPF after 8 weeks' treatment with BDP/F/G on markers of peripheral airway abnormalities or loss of elastic recoil in the parenchyma. | 8 weeks (4 weeks from V1 to V2; 4 weeks from V2 to V3)
  Improvement Δ1and Δ2 in Resonant Frequency (Hz) assessed by means of Impulse Oscillometry System (IOS).
To evaluate the effect of the increase of CPF after 8 weeks' treatment with BDP/F/G on respiratory symptoms and the perceived respiratory disability. | 8 weeks (4 weeks from V1 to V2; 4 weeks from V2 to V3)
  Improvement Δ1and Δ2 in dyspnoea perception assessed by modified Medical Research Council scale (mMRC) score. It is a five-point questionnaire (from 0 to 4) to assess the daily living activity-related breathlessness. Higher scores meaning a better outcome. COPD patients are considered at increased risk when their mMRC values are greater than 2.
To evaluate the effect of the increase of CPF after 8 weeks' treatment with BDP/F/G on quality of life. | 8 weeks (4 weeks from V1 to V2; 4 weeks from V2 to V3)
  Improvement Δ1 and Δ2 in COPD Assessment Test (CAT) score. It is a self-administered questionnaire consisting of eight items, which evaluate the most burdensome symptoms and limitations of the patients. The score for each item ranges from 0 to 5 and the total score (0 - 40) provides a simple and quantified measure of health-related quality of life, with higher scores indicating poorer health status. COPD patients are considered at increased risk when their CAT values are greater than 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine and Surgery, Respiratory Disease and Lung Function Unit, University of Parma, Italy, Parma, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected in a dedicated electronic Clinical Records Form (CRF). The database will be saved on a password- protected company personal computer which will be updated at each visit and used exclusively for scientific research purposes. At the time of enrolment, each patient will receive an alphanumeric code so that any information collected during the study, and in particular sensitive data, will be treated in an anonymous manner. Data reporting patients' identifications will only be used to file patients and collect informed consent.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Data will be available during the course of the study. The Investigator will keep paper and electronic copies of all documentation at the Center for a period of at least 7 years after the completion of the study and then he will arrange for its destruction.
Access Criteria: Only the personal delegated to collaborate with this study will be able to access to the database using a password to login.

REFERENCES:
- [Result] Rabe KF, Hurd S, Anzueto A, Barnes PJ, Buist SA, Calverley P, Fukuchi Y, Jenkins C, Rodriguez-Roisin R, van Weel C, Zielinski J; Global Initiative for Chronic Obstructive Lung Disease. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2007 Sep 15;176(6):532-55. doi: 10.1164/rccm.200703-456SO. Epub 2007 May 16. PMID 17507545
- [Result] Dal Vecchio L, Polese G, Poggi R, Rossi A. "Intrinsic" positive end-expiratory pressure in stable patients with chronic obstructive pulmonary disease. Eur Respir J. 1990 Jan;3(1):74-80. PMID 2178961
- [Result] Hellebrandova L, Chlumsky J, Vostatek P, Novak D, Ryznarova Z, Bunc V. Airflow limitation is accompanied by diaphragm dysfunction. Physiol Res. 2016 Jul 18;65(3):469-79. doi: 10.33549/physiolres.933064. Epub 2016 Apr 12. PMID 27070746
- [Result] Smith JA, Aliverti A, Quaranta M, McGuinness K, Kelsall A, Earis J, Calverley PM. Chest wall dynamics during voluntary and induced cough in healthy volunteers. J Physiol. 2012 Feb 1;590(3):563-74. doi: 10.1113/jphysiol.2011.213157. Epub 2011 Dec 5. PMID 22144580
- [Result] Sivasothy P, Brown L, Smith IE, Shneerson JM. Effect of manually assisted cough and mechanical insufflation on cough flow of normal subjects, patients with chronic obstructive pulmonary disease (COPD), and patients with respiratory muscle weakness. Thorax. 2001 Jun;56(6):438-44. doi: 10.1136/thorax.56.6.438. PMID 11359958
- [Result] Dean J, Panainte C, Khan N, Singh D. The TRIFLOW study: a randomised, cross-over study evaluating the effects of extrafine beclometasone/formoterol/glycopyrronium on gas trapping in COPD. Respir Res. 2020 Dec 9;21(1):323. doi: 10.1186/s12931-020-01589-5. PMID 33298062
- [Result] Singh D, Corradi M, Spinola M, Papi A, Usmani OS, Scuri M, Petruzzelli S, Vestbo J. Triple therapy in COPD: new evidence with the extrafine fixed combination of beclomethasone dipropionate, formoterol fumarate, and glycopyrronium bromide. Int J Chron Obstruct Pulmon Dis. 2017 Oct 6;12:2917-2928. doi: 10.2147/COPD.S146822. eCollection 2017. PMID 29062229
- [Result] French CL, Irwin RS, Curley FJ, Krikorian CJ. Impact of chronic cough on quality of life. Arch Intern Med. 1998 Aug 10-24;158(15):1657-61. doi: 10.1001/archinte.158.15.1657. PMID 9701100
- [Result] Vestbo J, Hurd SS, Agusti AG, Jones PW, Vogelmeier C, Anzueto A, Barnes PJ, Fabbri LM, Martinez FJ, Nishimura M, Stockley RA, Sin DD, Rodriguez-Roisin R. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2013 Feb 15;187(4):347-65. doi: 10.1164/rccm.201204-0596PP. Epub 2012 Aug 9. PMID 22878278
- [Result] Rogliani P, Matera MG, Facciolo F, Page C, Cazzola M, Calzetta L. Beclomethasone dipropionate, formoterol fumarate and glycopyrronium bromide: Synergy of triple combination therapy on human airway smooth muscle ex vivo. Br J Pharmacol. 2020 Mar;177(5):1150-1163. doi: 10.1111/bph.14909. Epub 2020 Jan 29. PMID 31660611
- [Result] Calzetta L, Cazzola M, Matera MG, Rogliani P. Adding a LAMA to ICS/LABA Therapy: A Meta-analysis of Triple Combination Therapy in COPD. Chest. 2019 Apr;155(4):758-770. doi: 10.1016/j.chest.2018.12.016. Epub 2019 Jan 17. PMID 30660781
- [Result] Cazzola M, Di Marco F, Santus P, Boveri B, Verga M, Matera MG, Centanni S. The pharmacodynamic effects of single inhaled doses of formoterol, tiotropium and their combination in patients with COPD. Pulm Pharmacol Ther. 2004;17(1):35-9. doi: 10.1016/j.pupt.2003.09.001. PMID 14643169
- [Result] Bestall JC, Paul EA, Garrod R, Garnham R, Jones PW, Wedzicha JA. Usefulness of the Medical Research Council (MRC) dyspnoea scale as a measure of disability in patients with chronic obstructive pulmonary disease. Thorax. 1999 Jul;54(7):581-6. doi: 10.1136/thx.54.7.581. PMID 10377201
- [Result] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809